CLINICAL TRIAL: NCT02379975
Title: Evaluation of Non-surgical Periodontal Therapy in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAIO VINICIUS GONÇALVES ROMAN TORRES (Other)
Responsible Party: Sponsor-Investigator, CAIO VINICIUS GONÇALVES ROMAN TORRES, PhD in Periodontology, Universidade Metropolitana de Santos
Organization: Universidade Metropolitana de Santos (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SantosMU 01
Record Dates: First submitted 2015-02-07; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis; Periodontitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rheumatoid arthristis (Experimental): individuals with rheumatoid arthritis
  Interventions: Procedure: Non-surgical Periodontal Therapy
- health (Active Comparator): healthy individuals
  Interventions: Procedure: Non-surgical Periodontal Therapy

INTERVENTIONS:
Procedure: Non-surgical Periodontal Therapy
  Other Names: periodontal scaling

SUMMARY:
Some clinical and epidemiological studies have revealed a high prevalence of periodontitis and tooth loss in patients with rheumatoid arthritis. The aim of this study was to evaluate the efficacy of periodontal scaling and oral hygiene instruction for patients with mild chronic periodontitis and rheumatoid arthritis through clinical periodontal parameters and laboratory tests for CRP (C- reactive protein) and ESR (erythrocyte sedimentation rate).

DETAILED DESCRIPTION:
This longitudinal study was approved by the Research Committee of the Santos Metropolitan University, and all individuals had access to the terms of consent. A total of 56 individuals with rheumatoid arthritis were assessed, and the investigators selected 12 women with a mean age of 45.38 who had been diagnosed with rheumatoid arthritis (RA) and who also had mild chronic periodontitis (PD). All of the patients were referred from the outpatient specialty medicals service and the rheumatologist's specialty outpatient clinic of the Metropolitan University of Santos diagnosed and evaluated individuals in the test group and the control group. The control group was composed of individuals who initiated periodontal treatment, did not have any systemic involvement, and had probing depth compatible with the individuals in the test group. The criteria for participation in the study included not having any dental procedure performed in the last six months, not having used antibiotic medication in the last six months, except for the use of drugs that could alter salivary flow (antidepressants, anxiolytics, antihistamines, and diuretics among others), not smoking, and not wearing braces.

The main parameters for the diagnosis of RA include counting the number of painful joints and the number of swollen joints, inflammatory activity (ESR and PCR), assessment of pain intensity, and assessment of joint mobility and functional capacity. Before the start of periodontal treatment, these tests were performed, and blood tests (ESR and PCR) were requested and evaluated by the rheumatologist in charge. The healthy subjects (control group) also underwent blood tests.

Upon completion of amamneses, periodontal clinical examinations were performed by a previously trained and calibrated periodontist, and in the sample studied, 10% were examined twice for each of the clinical criteria in order to obtain the intra-examiner reliability as measured by Kappa statistics (0.87).

The investigators observed the clinical parameters of periodontal probing depth (PD) in six points per tooth, and plaque index (PI) and gingival index (GI), conducted dichotomously for cheeks, buccal, mesial, distal and lingual/ palatal. All of the participants received radiographic, periapical, dental examinations in order to check the height level of the cortical bone.

Subjects received oral hygiene devices and underwent therapy for full mouth disinfection, and patients followed the protocol of holding two sessions with an interval of less than 24 hours between sessions. At the beginning of each session, oral hygiene instructions were given to each subject individually and the investigators tried to teach patients the correct way of using a brush and floss. The treatment was performed by scraping by a single periodontist who was blinded to the participants and the data obtained in clinical trials.

Each participant received seven doses of the individually-based mouthwash chlorhexidine 0.12%, to be used within seven calendar days after execution of the first session of the proposed therapy, and patients were told to always use it after brushing the last thing at night and then to wait 30 minutes to receive the maximum effectiveness of the chlorhexidine. After the procedures for dental scaling and root planing, 90 days passed before reassessment and new periodontal clinical and laboratory (ESR and PCR) tests were performed. Then the participants were referred to clinics operating in the college of Dentistry UNIMES as needed.

After tabulating the clinical and laboratory data for the participants included in this study, the data were subjected to statistical analysis. For this, the investigator used the software SPSS 13.0 and 5.0 bioestat. In all analytical situations a significance level of 95% should be adopted (α ≤.05). For each cluster of analytical interest, the characteristic distribution of the sample was tested and among the selected statistical tests being used were the statistical tests ANOVA with two factors (factor "health condition" - healthy or rheumatoid factor and "periodontal treatment" - Immediate evaluation or after periodontal treatment) and the Tukey's test.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* in control group, probing depth compatible with the individuals in the test group

Exclusion Criteria:

* not having any dental procedure performed in the last six months,
* not having used antibiotic medication in the last six months,
* except for the use of drugs that could alter salivary flow (antidepressants, anxiolytics, antihistamines, and diuretics among others),
* not smoking,
* and not wearing braces.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
periodontal probing depth (PD) | 90 days after periodontal therapy

SECONDARY OUTCOMES:
plaque index (PI) | 90 days after periodontal therapy
gingival index (GI) | 90 days after periodontal therapy
blood test erythrocyte sedimentation rate (ESR) | 90 days after periodontal therapy
blood test C-reactive protein (CRP) | 90 days after periodontal therapy

REFERENCES:
- [Background] Payne JB, Golub LM, Thiele GM, Mikuls TR. The Link Between Periodontitis and Rheumatoid Arthritis: A Periodontist's Perspective. Curr Oral Health Rep. 2015;2(1):20-29. doi: 10.1007/s40496-014-0040-9. PMID 25657894
- [Background] Olsen I, Potempa J. Strategies for the inhibition of gingipains for the potential treatment of periodontitis and associated systemic diseases. J Oral Microbiol. 2014 Aug 18;6. doi: 10.3402/jom.v6.24800. eCollection 2014. PMID 25206939
- [Background] Mikuls TR, Payne JB, Yu F, Thiele GM, Reynolds RJ, Cannon GW, Markt J, McGowan D, Kerr GS, Redman RS, Reimold A, Griffiths G, Beatty M, Gonzalez SM, Bergman DA, Hamilton BC 3rd, Erickson AR, Sokolove J, Robinson WH, Walker C, Chandad F, O'Dell JR. Periodontitis and Porphyromonas gingivalis in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 May;66(5):1090-100. doi: 10.1002/art.38348. PMID 24782175